CLINICAL TRIAL: NCT05791305
Title: Double Duty Interventions and Its Impact on DBM Among Children Under Five Years Ethiopia: A Cluster Randomized Controlled Trial
Brief Title: Double Duty Interventions and Its Impact on Double Burden of Malnutrition in Children Under Five Years
Acronym: DBM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Debre Berhan University (Other)
Responsible Party: Principal Investigator, Lemma Getacher, Principal investigator, Debre Berhan University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: DBU1112
Record Dates: First submitted 2023-03-06; First posted 2023-03-30 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Malnutrition; Malnutrition, Child; Obesity; Undernutrition; Thinness
Keywords: Double burden of malnutrition; Double-duty interventions; Children under five years; Undernutrition; Overnutrition
MeSH Terms: conditions — Malnutrition; Child Nutrition Disorders; Obesity; Thinness; Overnutrition

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial will be used.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): Will be provided an intervention.
  Interventions: Behavioral: double duty intervention packages
- Controll arm (No Intervention): Will not be provided the intervention.

INTERVENTIONS:
Behavioral: double duty intervention packages — The intervention employed in this study will serve as double-duty interventions. The WHO policy short report from 2017 and Hawkes et al2020 .'s were amended and used as the basis for the DDIs packages. The main components of the intervention packages are the promotion of a minimum level of dietary diversity, avoiding unwarranted harm from high-energy foods, and controlling market foods from the perspective of the consumer. The following central criteria will be used to evaluate the study's intervention packages.
  Arms: Intervention arm

SUMMARY:
Background: Double burden of malnutrition is an emerging public health problem among children under-five years due to the inevitable consequences of nutritional transition. Addressing these two contrasting forms of malnutrition (undernutrition and overnutrition) simultaneously brings an enormous challenge to the food and nutrition policies of developing countries like Ethiopia. Children under five ages are more vulnerable to DBM, especially during the first year of their life due to high growth and inadequate diet. Hence, there has been a paradigm shift in thinking to reduce its effect on the health of children. However, interventions that are used to address these different kinds of malnutrition are implemented through different governance and still, they are isolated and disintegrated each other. Therefore, double-duty interventions can tackle the risk of both nutritional problems simultaneously in an integrated approach through nutrition behavior change communication.

Objective: Therefore, the main aim of this pilot study is to assess the effect of selected double-duty interventions on the double burden of malnutrition among children under five years in Debre Berhan City, Ethiopia.

DETAILED DESCRIPTION:
Background: Double burden of malnutrition is an emerging public health problem among children under-five years due to the inevitable consequences of nutritional transition. Addressing these two contrasting forms of malnutrition (undernutrition and overnutrition) simultaneously brings an enormous challenge to the food and nutrition policies of developing countries like Ethiopia. Children under five ages are more vulnerable to DBM, especially during the first year of their life due to high growth and inadequate diet. Hence, there has been a paradigm shift in thinking to reduce its effect on the health of children. However, interventions that are used to address these different kinds of malnutrition are implemented through different governance and still, they are isolated and disintegrated each other. Therefore, double-duty interventions can tackle the risk of both nutritional problems simultaneously in an integrated approach through nutrition behavior change communication.

Objective: Therefore, the main aim of this pilot study is to assess the effect of selected double-duty interventions on the double burden of malnutrition among children under five years in Debre Berhan City, Ethiopia.

Methods: A cluster randomized controlled trial will be conducted among 456 under-five children (228 for each group) from January 25, 2023 to December 30, 2023. This pilot study will be used a one-year two-arm parallel cluster randomized controlled trial using clusters as a unit of randomization.

Expected outcomes: The endpoints expected from this pilot study are decreased double burden of malnutrition, improved minimum dietary diversity score, and decreased frequency of morbidity among children using double-duty interventions in the study area.

ELIGIBILITY:
Inclusion Criteria:

* who attend the intervention

Exclusion Criteria:

* who are not attended the intervention

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 456 (Estimated)
Dates: Start 2023-04-10 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of Double burden of malnutrition | 10 months
  Number of Mother of children who received double-duty interventions to reduce the DBM of children
Proportion of dietary diversity score | 10 months
  Number of Mother of children who received double-duty interventions to improve the dietary diversity score of children.
Proportion of low frequency of morbidity | 10 months
  Number of Mother of children who received double-duty interventions on the frequency of morbidity in children.

SECONDARY OUTCOMES:
Proportions of mothers with good maternal nutritional status | 10 months
  Proportions of mothers with good maternal nutritional status through questionnaire

CONTACTS AND LOCATIONS:
Locations (2):
- Ethiopia (2):
  - Debre Berhan University, Addis Ababa, Amhara
  - Health, Debre Berhan, Amhara

IPD SHARING:
Plan to Share IPD: No
This is a continued project.